CLINICAL TRIAL: NCT00411177
Title: Comparison of Post-dilution On-line Hemodiafiltration and Hemodialysis (TURKISH HDF STUDY)
Brief Title: Comparison of Post-dilution On-line Hemodiafiltration and Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ercan OK (Other)
Collaborators: Fresenius Medical Care North America (Industry)
Responsible Party: Sponsor-Investigator, Ercan OK, professor, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ege0683
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: End-Stage Renal Disease
Keywords: end-stage renal disease; hemodialysis; cardiovascular morbidity and mortality; high flux dialyser; on-line hemodiafiltration; arterial stiffness; inflammation; life quality; left ventricular hypertrophy
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation; Hypertrophy, Left Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Post-dilution on-line hemodiafiltration (Active Comparator): Post-dilution on-line hemodiafiltration
  Interventions: Procedure: post-dilution on-line hemodiafiltration
- High-flux hemodialysis (Other): High-flux hemodialysis
  Interventions: Procedure: high flux hemodialysis

INTERVENTIONS:
Procedure: post-dilution on-line hemodiafiltration — post-dilution on-line hemodiafiltration, 3 times a week 4 hours
  Arms: Post-dilution on-line hemodiafiltration
Procedure: high flux hemodialysis — High-flux hemodialysis, 3 times a week 4 hours
  Other Names: High-flux hemodialysis
  Arms: High-flux hemodialysis

SUMMARY:
This study aims to compare high-efficiency post-dilution on-line hemodiafiltration and high-flux hemodialysis regarding mortality, hospitalization rate, several clinical and laboratory parameters, and required medications.

The investigators hypothesize that high-efficiency post-dilution on-line hemodiafiltration may provide better outcome, less morbidity, higher quality of life, and lesser requirement of medications.

DETAILED DESCRIPTION:
The proposed controlled, randomized study aims to compare high-efficiency post-dilution on-line hemodiafiltration and high-flux hemodialysis regarding mortality, hospitalization rate, several clinical and laboratory parameters, and required medications.

Seven hundred and eighty HD patients will be taken into the study. The study will last for two years with an intermediate analysis at the first year. The patients will be randomly placed in two groups:

1. Post-dilution on-line hemodiafiltration,
2. High-flux hemodialysis.

In both groups, FX series high-flux helixone membranes will be used, duration of each session 240 minutes, and blood flow rates 250-400 ml/min. ONLINEplus integrated Fresenius 4008S machines will be used for on-line post-dilution HDF. Substitution volume will be above 15 liters in hemodiafiltration sessions.

Echocardiography for determination of left ventricular geometry, pulse wave velocity analysis to assess arterial stiffness, evaluation of nutritional and inflammatory state, assessment of life quality, depression and cost analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* on maintenance bicarbonate HD scheduled thrice weekly 12 hours/week,achieved mean single pool Kt/V above 1.2
* willingness to participate in the study with a written informed consent

Exclusion Criteria:

* To be scheduled for living donor renal transplantation
* To have serious life-limiting co-morbid situations, namely active malignancy, active infection, end-stage cardiac, pulmonary, or hepatic disease
* Pregnancy or lactating
* Current requirement for HD more than three times per week due to medical comorbidity
* GFR greater than 10 ml/min/1.73 m2 as measured by the average of urea and creatinine clearances obtained from a urine collection of at least 24 hours
* Use of temporary catheter
* Insufficient vascular access (blood flow rate lower than 250 ml/min)
* Mental incompetence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 782 (Actual)
Dates: Start 2007-01; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
composite of overall mortality and new cardiovascular events to include myocardial infarction, stroke, revascularization, and unstable angina pectoris requiring hospitalization. | two years

SECONDARY OUTCOMES:
cardiovascular mortality | two years
hospitalization rate | two years
intradialytic complications including hypotension and cramp | two years
health-related quality of life, depression burden, cognitive function | two years
required medications | two years
changes in blood pressure, left ventricular geometry, arterial stiffness, post-dialysis body weight, upper mid-arm circumference, hematocrit and related rHu-EPO doses, the levels of phosphorus, albumin, lipid parameters, hsCRP, and β-2 microglobulin | two years
postdialysis total body water determined by bioimpedance analysis | two years

CONTACTS AND LOCATIONS:
Overall Officials: Ercan Ok, MD, Principal Investigator — Ege University
Locations (2):
- Turkey (Türkiye) (2):
  - Ege University School of Medicine, Bornova, İzmir
  - FMC Clinics Turkey, Adana